CLINICAL TRIAL: NCT02318667
Title: An Open Label, Single Group Assignment Design Study to Correlate Soluble ST2 With Clinical, Endoscopic and Histological Activity in Moderate to Severe Ulcerative Colitis Patients Under Golimumab.
Brief Title: Correlation of Soluble Suppression of Tumorigenicity 2 (ST2) With Golimumab (MK-8259) Response in Participants With Ulcerative Colitis (UC) (MK-8529-022).
Acronym: EVOLUTION
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8259-022; 2014-003262-25 (EudraCT Number); MK-8259-022 (Other: Merck Protocol Number)
Record Dates: First submitted 2014-12-12; First posted 2014-12-17 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Colitis, Ulcerative
MeSH Terms: conditions — Colitis, Ulcerative | interventions — golimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Golimumab treatment (Experimental): Golimumab 200 mg initially administered by subcutaneous (SC) injection at Week 0, followed by 100 mg at Week 2 and then 50 mg or 100 mg every 4 weeks (per prescribing information) up to 16 weeks.
  Interventions: Biological: Golimumab

INTERVENTIONS:
Biological: Golimumab — Golimumab 50mg/0.5 mL in a single-use, ready-to-use autoinjector. Golimumab is a fully human anti-TNF (tumor necrosis factor) alpha monoclonal antibody that will be administered SC.
  Other Names: SIMPONI

SUMMARY:
The purpose of this study is to evaluate serum soluble human ST2 protein, the receptor for Interleukin-33 (IL-33) and a member of the proinflammatory Interleukin-1 (IL-1) receptor superfamily, as a surrogate biological marker predictive of disease outcome and therapeutic response to golimumab treatment in participants with moderate to severe UC who have failed on prior conventional therapies. The primary endpoints of this study are to correlate serum soluble ST2 levels with endoscopic activity (endoscopic subscore of the Mayo score) and histological activity (Geboes index) of disease.

ELIGIBILITY:
Inclusion Criteria:

* Inadequate response to conventional therapy including corticosteroids or are intolerant to, or have medical contraindications for conventional therapies
* UC diagnosed prior to screening, based on a biopsy collected at endoscopy
* Moderate to severe active UC with total Mayo score of 6 to 12, inclusive at baseline, and endoscopic Mayo sub-score, greater than or equal to 2
* Adenomatous polyps removed within last 5 years or at the screening visit prior to the first drug treatment
* Extensive colitis for ≥ 8 years, or disease limited to the left side of the colon for ≥10 years should have a colonoscopy to exclude the presence of dysplasia within 1 year prior to study inclusion or a colonoscopy to exclude the presence of malignancy at the screening visit
* No history of untreated latent or active Tuberculosis (TB) prior to screening
* Negative stool results for enteric pathogens

Exclusion Criteria:

* History of asthma
* History of autoimmune diseases
* History of hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-02-27 (Actual); Primary Completion 2017-06-21 (Actual); Study Completion 2017-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Magro F, Lopes S, Silva M, Coelho R, Portela F, Branquinho D, Correia L, Fernandes S, Cravo M, Caldeira P, Sousa HT, Patita M, Lago P, Ramos J, Afonso J, Redondo I, Machado P, Cornillie F, Lopes J, Carneiro F; Portuguese IBD Group [GEDII]. Low Golimumab Trough Levels at Week 6 Are Associated With Poor Clinical, Endoscopic and Histological Outcomes in Ulcerative Colitis Patients: Pharmacokinetic and Pharmacodynamic Sub-analysis of the Evolution Study. J Crohns Colitis. 2019 Oct 28;13(11):1387-1393. doi: 10.1093/ecco-jcc/jjz071. PMID 30989180
- [Result] Magro F, Lopes S, Silva M, Coelho R, Portela F, Branquinho D, Correia L, Fernandes S, Cravo M, Caldeira P, Tavares de Sousa H, Patita M, Lago P, Ramos J, Afonso J, Redondo I, Machado P, Philip G, Lopes J, Carneiro F. Soluble human Suppression of Tumorigenicity 2 is associated with endoscopic activity in patients with moderate-to-severe ulcerative colitis treated with golimumab. Therap Adv Gastroenterol. 2019 Aug 30;12:1756284819869141. doi: 10.1177/1756284819869141. eCollection 2019. PMID 31516554

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Golimumab Treatment
Started | 38
Completed | 29
Not Completed | 9
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 6
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 38
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.8 (12.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Serum human Suppression of Tumorigenicity 2 (ST2) level [Mean (Standard Deviation); unit: ng/mL] — ST2, a serum biomarker, was collected at Baseline. Population: Participants with available ST2 data
  ng/mL
    number analyzed (Participants) | 34
    (all) | 21.8 (11.09)

OUTCOME MEASURES:

1. Primary Outcome: Serum ST2 Level at Week 6
Description: ST2, a serum biomarker, was collected at Week 6. ST2 levels were used to determine whether or not there is a correlation with endoscopic or histologic activity, or a clinical response to treatment in participants with moderate to severe Ulcerative Colitis.
Time Frame: Week 6
Population: Participants with available Week 6 ST2 data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 34
ng/mL | 21.8 (14.41)

2. Primary Outcome: Correlation of Serum Soluble ST2 Levels With Endoscopic Activity of Disease (Assessed by Endoscopy Subscore of Mayo Score) at Week 6
Description: ST2, a serum biomarker, was collected at Week 6. Endoscopic Mayo subscore is one of 4 components that comprise the total Mayo Score, a scale for assessing ulcerative colitis (UC) activity. Endoscopic Mayo subscore ranges from 0-3: 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern, mild friability); 2 = moderate disease (marked erythema, absent vascular pattern, friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration). A higher score indicates more severe disease. Moderate correlation was defined as a Spearman correlation (rs) coefficient between -0.5 to -0.3 or 0.3 to 0.5.
Time Frame: Week 6
Population: Analysis population includes all participants who had received study medication, had at least one valid post-baseline assessment for the primary endpoint that correlates ST2 with endoscopic activity and/or histological activity, and had a Week 6 endoscopic Mayo subscore.
Measure: Number (95% Confidence Interval); unit: Spearman correlation (rs) coefficient
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 34
Spearman correlation (rs) coefficient | 0.451 [0.133 to 0.685]
Statistical Analysis 1: Comparison: Golimumab Treatment; Test type: Other; p = 0.0074, t-test, 2 sided

3. Primary Outcome: Correlation of Serum Soluble ST2 Levels With Histological Activity (Assessed by Geboes Index) at Week 6
Description: ST2, a serum biomarker, was collected at Week 6. Geboes index, is a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher score indicates more severe disease. Moderate correlation was defined as rs coefficient between -0.5 to -0.3 or 0.3 to 0.5.
Time Frame: Week 6
Population: Analysis population includes all participants who had received study medication, had at least one valid post-baseline assessment for the primary endpoint that correlates ST2 with endoscopic activity and/or histological activity, and had a Week 6 Geboes index score.
Measure: Number (95% Confidence Interval); unit: rs coefficient
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 34
rs coefficient | 0.252 [-0.094 to 0.544]
Statistical Analysis 1: Comparison: Golimumab Treatment; Test type: Other; p = 0.1506, t-test, 2 sided

4. Secondary Outcome: Serum ST2 Level at Week 16
Description: ST2, a serum biomarker, was collected at Week 16. ST2 levels were used to determine whether or not there is a correlation with endoscopic or histologic activity, or a clinical response to treatment in participants with moderate to severe Ulcerative Colitis.
Time Frame: Week 16
Population: Participants with available Week 16 ST2 data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 29
ng/mL | 17.9 (13.10)

5. Secondary Outcome: Correlation of Serum Soluble ST2 Levels With Endoscopic Activity (Assessed by Endoscopy Subscore of Mayo Score) at Week 16
Description: ST2, a serum biomarker, was collected at Week 16. Endoscopic Mayo subscore is one of 4 components that comprise the total Mayo Score, a scale for assessing ulcerative colitis (UC) activity. Endoscopic Mayo subscore ranges from 0-3: 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern, mild friability); 2 = moderate disease (marked erythema, absent vascular pattern, friability, erosions); 3 = Severe disease (spontaneous bleeding, ulceration). A higher score indicates more severe disease. Moderate correlation was defined as rs coefficient between -0.5 to -0.3 or 0.3 to 0.5.
Time Frame: Week 16
Population: Analysis population includes all participants who had received study medication and had at least one valid post-baseline assessment for the primary endpoint that correlates ST2 with endoscopic activity and/or histological activity, and had a Week 16 endoscopic Mayo subscore.
Measure: Number (95% Confidence Interval); unit: rs coefficient
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 29
rs coefficient | 0.268 [-0.109 to 0.578]

6. Secondary Outcome: Correlation of Serum Soluble ST2 Levels With Histological Activity (Assessed by Geboes Index) at Week 16
Description: ST2, a serum biomarker, was collected at Week 16. Geboes index, is a validated score for evaluating histologic disease activity in UC as follows: grade 0 = structural and architectural changes; grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher score indicates more severe disease. Moderate correlation was defined as rs coefficient between -0.5 to -0.3 or 0.3 to 0.5.
Time Frame: Week 16
Population: Analysis population includes all participants who had received study medication and had at least one valid post-baseline assessment for the primary endpoint that correlates ST2 with endoscopic activity and/or histological activity, and had a Week 16 Geboes index score.
Measure: Number (95% Confidence Interval); unit: rs coefficient
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 29
rs coefficient | 0.177 [-0.202 to 0.511]

7. Secondary Outcome: Correlation of Serum Soluble ST2 Levels With Faecal Calprotectin Levels at Baseline and Week 6 and Week 16
Description: ST2 and faecal calprotectin, serum biomarkers, were collected at Week 6 and Week 16. Faecal calprotectin is a surrogate marker for the presence of intestinal inflammation and response to treatment in participants with Inflammatory Bowel Disease. Moderate correlation was defined as rs coefficient between -0.5 to -0.3 or 0.3 to 0.5.
Time Frame: Baseline, Weeks 6 and 16
Population: Analysis population includes all participants who had received study medication and had a valid faecal calprotectin assessment at time point (Baseline, Week 6, and Week 16).
Measure: Number (95% Confidence Interval); unit: rs coefficient
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 32
rs coefficient
  Baseline | 0.146 [-0.214 to 0.470]
  Week 6: number analyzed (Participants) | 31
  Week 6 | -0.022 [-0.374 to 0.335]
  Week 16: number analyzed (Participants) | 28
  Week 16 | -0.140 [-0.487 to 0.246]

8. Secondary Outcome: Correlation of Serum Soluble ST2 Levels With Clinical Activity (Assessed by Total Mayo Score) at Week 6 and Week 16
Description: ST2, a serum biomarker, was collected at Week 6 and Week 16. The total Mayo Score, is a scale for assessing UC activity and is the sum of 4 subscores (assessment of stool frequency [0-3], rectal bleeding [0-3], Physician's Global Assessment [0-3], and endoscopic Mayo subscore [0-3]) and has values that range from 0 to 12. Clinical remission: ≤2 points with no individual subscore > 1; Mildly active disease: 3-5 points; Moderately active disease: 6-10 points; Severely active disease: 11-12 points. A higher score indicates more severe disease. Moderate correlation was defined as rs coefficient between -0.5 to -0.3 or 0.3 to 0.5.
Time Frame: Weeks 6 and 16
Population: Analysis population includes all participants who had received study medication and had at least one valid post-baseline assessment for the primary endpoint that correlates ST2 with endoscopic activity and/or histological activity, and total Mayo score at Weeks 6 and 16.
Measure: Number (95% Confidence Interval); unit: rs coefficient
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 34
rs coefficient
  Week 6 | 0.404 [0.076 to 0.653]
  Week 16: number analyzed (Participants) | 29
  Week 16 | 0.098 [-0.279 to 0.448]

9. Secondary Outcome: Change From Baseline to Week 6 in ST2 Levels in Participants With Active Versus Inactive UC
Description: ST2, a serum biomarker, was collected at Baseline and Week 6. Active Ulcerative Colitis was defined as an endoscopic Mayo subscore ≥2 and inactive Ulcerative Colitis was defined as an endoscopic Mayo subscore of 0 or 1.
Time Frame: Baseline, Week 6
Population: Analysis population includes all participants who had received study medication and had at least one valid post-baseline assessment for the primary endpoint that correlates ST2 with endoscopic activity and/or histological activity at Week 6.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Inactive Disease: Participants with inactive Ulcerative Colitis at Week 6
- Active Disease: Participants with active Ulcerative Colitis at Week 6
Arm/Group | Inactive Disease | Active Disease
Number analyzed (Participants) | 14 | 20
ng/mL
  Baseline | 17.2 (6.81) | 25.0 (12.47)
  Change from baseline at Week 6 | -3.5 (6.89) | 2.4 (7.75)

10. Secondary Outcome: Change From Baseline to Week 6 in ST2 Level According to Participant's Mayo Endoscopic Response at Week 16 (Maintained Response at Week 16 or Did Not Maintain Response at Week 16)
Description: ST2, a serum biomarker, was collected at Baseline and Week 6. Comparison of participants who achieved endoscopic response [endoscopic Mayo subscore 0 or 1] at Week 6 and maintained response through Week 16 versus participants who did not maintain response throughout Week 16, regarding serum soluble ST2 at baseline, Week 6 and change between baseline and Week 6.
Time Frame: Baseline, Week 6
Population: Analysis population includes all participants who had received study medication and achieved endoscopic response at Week 6.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Maintained Endoscopic Response: Participants who achieved endoscopic response at Week 6 and maintained endoscopic response at Week 16
- Did Not Maintain Endoscopic Response: Participants who achieved endoscopic response at Week 6 and did not maintain endoscopic response at Week 16
Arm/Group | Maintained Endoscopic Response | Did Not Maintain Endoscopic Response
Number analyzed (Participants) | 10 | 4
ng/mL
  Baseline | 15.7 (6.06) | 21.0 (8.01)
  Change from Baseline at Week 6 | -1.8 (7.28) | -7.8 (3.68)

11. Secondary Outcome: Correlation of Endoscopic Mayo Subscore With Ulcerative Colitis Endoscopic Index Of Severity (UCEIS©) Overall Score at Week 6 and Week 16
Description: UCEIS© is a 3-item (vascular pattern, bleeding and erosion/ulceration) validated tool for assessing endoscopic severity of UC. Each item has 3 or 4 levels of severity and is given a score. The scores for each individual item are combined into a total score ranging from 1 to 11. A higher score indicates increased endoscopic severity of UC. Moderate correlation was defined as rs coefficient between -0.5 to -0.3 or 0.3 to 0.5.
Time Frame: Week 6 and Week 16
Population: Analysis population includes all participants who had received study medication and had at least one valid post-baseline assessment for the primary endpoint that correlates ST2 with endoscopic activity and/or histological activity, and UCEIS overall score at Week 6 and Week 16.
Measure: Number (95% Confidence Interval); unit: rs coefficient
Arm/Group | Golimumab Treatment
Number analyzed (Participants) | 34
rs coefficient
  Week 6 | 0.830 [0.683 to 0.912]
  Week 16: number analyzed (Participants) | 29
  Week 16 | 0.875 [0.748 to 0.940]

ADVERSE EVENTS:
Time Frame: Up to 16 weeks
Description: Analysis population includes all participants who received at least one dose of study medication.
Arm/Group | Golimumab Treatment
All-Cause Mortality (participants affected / at risk) | 0/38
Serious Adverse Events (participants affected / at risk) | 4/38
Other Adverse Events (participants affected / at risk) | 4/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab Treatment (N=38)
Colitis ulcerative (Gastrointestinal disorders) | 3 (4)
Pneumonia (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Golimumab Treatment (N=38)
Colitis ulcerative (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT02318667/Prot_SAP_000.pdf